CLINICAL TRIAL: NCT02161887
Title: The Healing Context in CAM: Instrument Development and Initial Validation - Phase 3 Validation Study
Brief Title: The Healing Context in Complementary and Alternative Medicine (CAM): Initial Validation Study
Acronym: HEAL
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Carol Greco, Assistant Professor of Psychiatry, University of Pittsburgh
Other Study IDs: AT006453-3
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Chronic Low Back Pain; Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Complementary Medicine Group: Patients receiving chiropractic care, acupuncture, or meditation for chronic pain
- Conventional Medicine Group: Patients receiving conventional medicine care (physical therapy, medication management) for chronic pain.

SUMMARY:
The overall objective of this study is to develop and test an efficient set of self-report instruments to measure Complementary and Alternative Medicine(CAM)-relevant contextual factors important in healing. The initial phase of the study involves developing and refining an item bank. During the initial 'item bank development' phase, the investigators will run focus groups and cognitive interviews with individuals who participate in CAM and conventional medicine interventions. The next step of instrument development is called Calibration, and involves administering the revised item bank to an internet sample and to persons who receive services in a CAM clinic and a conventional primary care setting. The items will be calibrated using item response theory and classical test theory. This will result in a computerized adaptive testing version of the instrument, as well as a static short form of the instrument. This current protocol in ClinicalTrials.gov pertains only to the final, Validation Phase of the study. The final phase of the project will involve conducting initial validation studies of the set of instruments. The set of instruments will be called the Healing Encounters and Attitudes Lists (HEAL). The investigators will evaluate the convergent, discriminant, and predictive validity of the HEAL instruments in a sample of 200 persons with chronic low back pain or neck pain who are receiving physical therapy, chiropractic care, acupuncture, medical management, or mindfulness-based stress reduction. For convergent validity, the HEAL is expected to display moderate to large correlations with measures of similar constructs. The HEAL is expected to correlate modestly with self-report measures of general psychosocial functioning, in support of discriminant validity. Finally, HEAL scores should account for a significant proportion of the variance in treatment outcome, supporting predictive validity.

DETAILED DESCRIPTION:
This project will develop and test a set of patient self-report measurement tools to assess the perceived contextual factors, such as patient attitudes and expectations, patient provider relationship factors, and environmental factors that contribute to healing. This project is synergistic with the National Institutes of Health (NIH) Roadmap initiative, Patient Reported Outcomes Measurement Information System (PROMIS), and will use the rigorous instrument development and validation methodology of PROMIS. The overall objective of this study is to develop efficient self-report instruments to measure CAM-relevant contextual factors important in healing, hereafter referred to as the Healing Encounters and Attitudes Lists (HEAL), and conduct initial validation in persons seeking CAM and conventional treatment for pain. Specific Aim 1: Develop item banks. The investigators will employ several iterative steps used successfully in PROMIS to identify items that assess contextual factors of healing relevant to CAM. Initial steps in developing item banks include: a) compilation and evaluation of existing instruments and relevant questions, b) consultation with experts, and c) focus groups with individuals who participate in CAM and conventional medicine interventions, and d) item editing. During the initial phase of this study, the investigators expect to identify conceptual areas of potential importance to CAM interventions and patients, and identify and edit items to create item banks assessing these conceptual areas. Specific Aim 2: Calibrate items. The investigators will use item response theory (IRT) and classical test theory (CTT) to calibrate the items from Aim 1 on three samples: 1) an internet-based sample (n= 1400), 2) 125 outpatients participating in CAM interventions at the Center for Integrative Medicine (CIM), and 3) 125 outpatients at a General Internal Medicine clinic. During year 3-4 the investigators will administer the items in the item banks to the 1650 persons, conduct IRT and CTT analyses and refine the item banks to only those items that best assess the constructs. Specific aim 2 will result in Computerized Adaptive Testing (CAT) versions of the HEAL, which maximizes information while minimizing patient time burden. Static short forms of the HEAL item banks will be derived from the HEAL CATs in Aim 2. Specific Aim 3: Conduct initial validation studies. The investigators will evaluate convergent, discriminant, and predictive validity of the Healing Encounters and Attitudes List (HEAL) in a sample of chronic low back pain (CLBP) or neck pain patients receiving CAM and conventional medicine treatments. The validity studies will use two samples of adults with CLBP: 100 persons receiving CAM treatments: chiropractic manipulation (CM), acupuncture, or mindfulness-based stress reduction (MBSR) at the CIM, and 100 persons receiving conventional care (physical therapy or medical management) at the University of Pittsburgh Medical Center (UPMC). The investigators will administer the CAT version of the HEAL questionnaire developed in aims 1 and 2 as well as conventional measures of treatment expectancy, confidence in treatment provider, psychosocial functioning, and pain and disability treatment outcome measures for CLBP and neck pain. • Hypothesis 3a: Scores on the HEAL measures will display moderate to large correlations (r's > .50) with similar self-report measures, supporting convergent validity. • Hypothesis 3b: Scores on the HEAL measures will correlate modestly (r's = .20-.35) with self-report measures of general psychosocial functioning, supporting discriminant validity. • Hypothesis 3c: HEAL scores will account for a significant proportion of variance in treatment outcome in both samples. In addition, the investigators predict that HEAL scores will demonstrate incremental validity, i.e., the scores will account for significant incremental variance in outcome beyond that accounted for by existing measures of treatment expectancy and related constructs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older; able to read and understand English; able to use a computer; starting a new treatment for back or neck pain, or started treatment within the past month.

Exclusion Criteria:

* psychotic disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are beginning or about to begin CAM or Conventional Medicine treatments for chronic back pain or chronic neck pain in Pittsburgh, Pennsylvania at University of Pittsburgh Medical Center (UPMC).
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression of Change (CGI) | 6 - 8 weeks, 4 months post study entry

SECONDARY OUTCOMES:
Roland and Morris Disability Questionnaire | Baseline, 6-8 weeks, 4 months post baseline

OTHER OUTCOMES:
Neck Disability Index | Baseline, 6-8 weeks, 4 months post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Carol M Greco, Ph.D., Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC General Clinical Research Center, Pittsburgh, Pennsylvania
  - UPMC Shadyside Center for Integrative Medicine, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Greco CM, Glick RM, Morone NE, Schneider MJ. Addressing the "It Is Just Placebo" Pitfall in CAM: Methodology of a Project to Develop Patient-Reported Measures of Nonspecific Factors in Healing. Evid Based Complement Alternat Med. 2013;2013:613797. doi: 10.1155/2013/613797. Epub 2013 Dec 19. PMID 24454501
- [Background] Greco CM, Yu L, Johnston KL, Dodds NE, Morone NE, Glick RM, Schneider MJ, Klem ML, McFarland CE, Lawrence S, Colditz J, Maihoefer CC, Jonas WB, Ryan ND, Pilkonis PA. Measuring nonspecific factors in treatment: item banks that assess the healthcare experience and attitudes from the patient's perspective. Qual Life Res. 2016 Jul;25(7):1625-34. doi: 10.1007/s11136-015-1178-1. Epub 2015 Nov 12. PMID 26563249